CLINICAL TRIAL: NCT00575211
Title: Genetic Modulation of Left Ventricular Recovery in Recent Onset Cardiomyopathy
Brief Title: Study Looking at the Recovery of New Onset Cardiomyopathy
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Dennis McNamara, Professor of Medicine, University of Pittsburgh
Other Study IDs: IMAC II; NIH grant
Record Dates: First submitted 2007-12-14; First posted 2007-12-18 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Cardiomyopathy
Keywords: New onset cardiomyopathy; Onset of symptoms less than 6 months; LVEF < 40%
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — At time of enrollment, 30cc of blood will be obtained: 10cc for plasma banking for neurohormones and cytokine analysis, 10 cc for DNA banking and genotyping, 5 cc for evaluation of gene expression of inflammatory markers from circulating leukocytes and 5 cc for serum banking. Ten ccs of blood for cytokine analysis will also be collected at one month and six months after entry. A blood specimen for repeat analysis of serum mediator (5ccs in a red top tube) will be drawn at six months and sent to the University of Pittsburgh. All blood samples will be kept for 10 years. Access to the banked DNA will be limited to investigations at the University of Pittsburgh and each site of this multi-center trial. These samples will be available without any identifying information (name, social security number and medical record number). In addition, a Certificate of Confidentiality has been obtained from the NIH for further subject protection.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cardiomyopathy

SUMMARY:
This is a multi-center, prospective evaluation of left ventricular recovery on conventional therapy in patients with the recent onset of dilated cardiomyopathy. In some subjects with this disorder, the heart will recover significantly over the first year, while others will be left with a chronically weak heart. The proteins that help the heart recover are encoded by genes, which can differ markedly between individuals. The goal of the current study is to determine whether variation in these genes involved affect the probability that the heart will recover. We will also look at which genes are involved in inflammation and which ones are "turned on" (producing proteins) in circulating white blood cells.{These statements will only be added if the site has chosen to participate in RNA analysis}. In addition, this study will look at how levels of proteins in the blood, proteins called "cytokines' which control inflammation and proteins called "neurohormones" which are released when the heart weakens, affect the likelihood of recovery.

Enrollment will take place at 15 centers. The goal is to enroll approximately 500 adult subjects (age 18 years or older, both men and women) over the course of approximately 48 months.

DETAILED DESCRIPTION:
After presenting with new onset idiopathic dilated cardiomyopathy, one third of patients experience dramatic recovery of left ventricular function, while for the majority chronic heart failure and left ventricular dysfunction persist. This marked variation in clinical outcomes is determined in part by genetic heterogeneity of the systemic response to myocardial injury. This population has been excluded from most clinical trials and few studies have examined the role of cytokine and neurohormonal mediators in modulating the balance between left ventricular recovery and remodeling in early cardiomyopathy. This proposal will investigate whether genetic polymorphisms of inflammatory and neurohormonal mediators influence subsequent clinical outcomes for patients with recent onset primary (idiopathic) dilated cardiomyopathy. The study will enroll 500 patients with recent onset left ventricular dysfunction (LVEF < 0.40) due to non-ischemic primary cardiomyopathy at eleven centers and follow these patients prospectively to evaluate subsequent left ventricular recovery and freedom from clinical events.

Specific aim 1 will be to determine the correlation of echocardiographic parameters of systolic and diastolic functional entry with circulating inflammatory mediators: TNF, IL-6 and TNF receptors 1 and 2. Specific aim 2 will be to determine the predictive value of early plasma TNFα levels and of left ventricular size by transthoracic echo at baseline in predicting improvements in left ventricular ejection function (LVEF) at 6 months. Specific aim 3 will evaluate the effects of the TNFA 1/2 promoter polymorphism on circulating plasma TNF levels and its influence on subsequent improvement in LVEF. Specific aim 4 will look at the impact of the deletion allele of the angiotensin-converting enzyme and the genetic variation of beta 1 and beta 2 adrenergic receptors on left ventricular recovery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 18 years or over, and may be of either gender and of any race.
2. Patients must have significantly systolic dysfunction, defined as a left ventricular ejection fraction of less than or equal to 40% by transthoracic echocardiography.
3. The patients must have a recent onset of dilated cardiomyopathy. Specifically, the initial signs or symptoms of cardiomyopathy should not pre-date the time of evaluation for the study by more than six months.
4. Subjects diagnosed during with peripartum cardiomyopathy (PPCM) are allowed as long as they are enrolled within six months of cardiac symptoms.
5. Subjects presenting with acute heart failure with a positive familial history of cardiomyopathy are included. Subjects who are asymptomatic, but are diagnosed with a cardiomyopathy of unknown duration during screening for known familial disease are excluded
6. Patients must be competent to give informed consent.

Exclusion Criteria:

1. Coronary artery disease as defined as a single coronary artery stenosis of a major epicardial vessel greater than 50% or a previous history of myocardial infarction.
2. Patients with a history of familial cardiomyopathy, or a primary relative defined as parents, siblings or children with a dilated cardiomyopathy are excluded.
3. Past or present history of alcoholism, or in whose current alcohol consumption exceeds an average of three drinks per day. A past history of cocaine or IV drug abuse as a possible explanation for their cardiomyopathy as well as substance abuse of prescription pain relievers or any illicit drug that may hinder the participant's ability to complete study follow-up.
4. Patients who are post cardiac transplant.
5. Patients whose heart failure is felt to be secondary to primary valvular disease, uncorrected thyroid disease, uncontrolled hypertension despite medical therapy, obstructive or hypertrophic cardiomyopathy, pericardial disease, or a systemic illness such as sarcoidosis.
6. Patients whose history of cardiac symptoms or signs of cardiac disease predate the time of evaluation by more than six months are excluded.
7. Evidence of ongoing bacteremia or sepsis. Patient with a febrile illness felt to be secondary to myocarditis can be included (even with a non-diagnostic biopsy) if a bacteriologic cause of the illness is excluded.
8. Patients with other life threatening diseases such as malignancy which would likely decrease their life expectancy over the next three years. Any history of malignancy treated with either chest radiation or chemotherapy.
9. The following patients are excluded for medical reasons: Patients with evidence of chronic liver disease (total bilirubin >3.0mg%) or chronic renal disease (creatinine > or equal to 2.5mg%) are excluded from the study. Subjects who present with an acute worsening of renal function or liver function tests in the setting of potentially fulminant myocarditis can be enrolled. Patients whose hepatic abnormalities are secondary to hypoperfusion can also be considered.
10. Patients with previous history of diabetes and with evidence of multisystem end organ damage (i.e. end stage renal disease and cardiomyopathy) or with evidence of any coronary disease. Patient with diabetes without significant end organ damage is allowed.
11. Patients enrolled in other placebo controlled experimental trials.
12. Patients who have had a myocardial biopsy, which reveals evidence of hemochromatosis, amyloid, sarcoidosis, or giant cell myocarditis, are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: New onset Cardiomyopathy patient with symptoms less than 6 months
Sampling Method: Non-Probability Sample
Enrollment: 373 (Actual)
Dates: Start 2004-01; Primary Completion 2010-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to determine whether variation in genetic background influences clinical outcomes in new onset cardiomyopathy. | 5 years

SECONDARY OUTCOMES:
Determine whether cytokine or echo parameters can predict who will have significant recovery left ventricular function. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Dennis McNamara, MD, Principal Investigator — University of Pittsburgh
Locations (16):
- United States (14):
  - University of California - Irvine, Orange, California
  - University of Florida, Gainesville, Florida
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - University of Rochester Medical Center, Rochester, New York
  - Wake Forest Univesity Health Sciences, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center, Dalls, Texas
  - The Methodist Hospital, Houston, Texas
- Canada (2):
  - University Health Network, Toronto, Ontario
  - SBMB Jewish General Hospital, Montreal, Quebec

REFERENCES:
- [Derived] McNamara DM, Starling RC, Cooper LT, Boehmer JP, Mather PJ, Janosko KM, Gorcsan J 3rd, Kip KE, Dec GW; IMAC Investigators. Clinical and demographic predictors of outcomes in recent onset dilated cardiomyopathy: results of the IMAC (Intervention in Myocarditis and Acute Cardiomyopathy)-2 study. J Am Coll Cardiol. 2011 Sep 6;58(11):1112-8. doi: 10.1016/j.jacc.2011.05.033. PMID 21884947